CLINICAL TRIAL: NCT03220659
Title: Optimising Pacemaker Therapy Using Multi-point Pacing (the OPT-MPP Study)
Acronym: OPT-MPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, KK Witte, Senior, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 229391
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard settings (Placebo Comparator): Usual pacing programming
  Interventions: Device: Standard settings
- Multi-point pacing (Experimental): MPP programming
  Interventions: Device: Multi-point pacing

INTERVENTIONS:
Device: Multi-point pacing — Pacing from more than one pole from the left ventricular lead
  Other Names: MPP
  Arms: Multi-point pacing
Device: Standard settings — Normal bipolar LV pacing
  Other Names: CRT pacing
  Arms: Standard settings

SUMMARY:
Recently, the introduction of quadripolar left ventricular leads (one with four pacing poles) has allowed the opportunity to pace the lateral (back) of the heart from several points at once using a single lead (multi-point pacing - MPP). Although it seems logical that electrical beginning at several points on the left ventricular wall should improve coordination of the heart, there is no consistent response in terms of improved remodeling (cardiac structure and function) or composite scores of patient-related status. The technology has a further disadvantage that it leads to accelerated battery drain, with on average one year less longevity over the lifetime of the device.

Aims are:

1. to explore the effect of MPP on the force-frequency relationship,
2. to examine the effects of MPP on exercise capacity measured by treadmill walk time and whether these are related to the FFR response to MPP in individual patients,
3. establish whether the acute contractile response is maintained to 6 months after the implant procedure and
4. determine whether the acute contractile response to MPP is associated with subsequent beneficial remodeling over a further six months.

DETAILED DESCRIPTION:
Cardiac function during exercise Cardiac output is a function of stroke volume (the volume of blood ejected with each beat) and heart rate. During exercise cardiac output must rise to supply exercising muscles. This occurs by an increase in both heart rate and stroke volume. Limitations to heart rate rise (chronotropic incompetence (CI)) or stroke volume increases (contractility) or a combination of both might contribute to lower cardiac output during exercise.

Increases in contractility during exercise are under two major influences: depolarization-rate dependent (heart rate dependent), and catecholamine-dependent. Normal increases in contractility during exercise require both to be functioning normally. As mentioned, the catecholamine system is chronically overactive in CHF such that there is down-regulation of receptors making the sympathetic system less sensitive and responsive. The depolarization-rate dependent (catecholamine-independent) mechanism, whereby increases in heart rate lead to increases in the force of contraction known as the Treppe phenomenon, or the force frequency relationship (FFR), was described by Bowditch in the late 19th century, and is thought to be impaired in CHF such that contractility in heart failure does not rise normally with increases in heart rate and in fact reduces once heart rate rises above a threshold.

How to determine force-frequency relationship in humans

The investigators have established a reliable, reproducible and non-invasive method by which to assess the FFR in patients with pacemaker devices. The investigators subsequently demonstrated that optimizing heart rate rise to within the range for optimal contractility is associated with acute improvements in exercise capacity. The FFR assessment protocol is described below.

This study will have two phases:

For the first stage, 50 patients undergoing cardiac resynchronisation therapy will be invited, to participate in an observational, double-blind, randomised cross-over study exploring the acute effects of multi-point pacing (MPP) on the force frequency relationship and exercise capacity at around 6 weeks and 6 months following the implant. The plan is not to explore whether MPP improves remodeling following a CRT implant so MPP will be programmed off during the first 6 months after implantation.

At the end of the first six months, if there are promising results from the first stage, participants will then randomly be allocated to MPP on or off in a double-blind parallel group study. After a further 6 months (12 months after the initial implant) they will return for a single visit during which they will have an echocardiogram and exercise test.

Six weeks following device implant (phase 1)

At the first visit, participants will undergo a pacemaker check, a review of medications and other medical history. They will sign a consent form. They will then undergo a resting echocardiogram.

Following this, their pacemaker will be randomly programmed to MPP or usual pacing. Programming will be performed by a secondary (unblinded) cardiac physiologist, who will also be responsible for watching the electrocardiogram during each test. Patients and the primary cardiac physiologist undertaking the echocardiogram will be unaware of allocation. Images will be collected at rest following which atrial pacing will be initiated in the DDD-mode at 50 beats/min (or the next highest 'round figure' above the baseline heart rate). After four minutes, images will be recorded, and the pacing rate will then be increased in a stepwise 20-beat interval with images recorded after every four minutes. This step-wise increase will be repeated until the maximum predicted heart rate as per the calculation by Astrand (220-age) is reached. At this point peak data will be collected and pacing will then return to baseline settings. Throughout this assessment, at each stage a blood pressure will be recorded to allow the calculation of the force frequency relationship. Five minutes after the end of atrial pacing, a final set of images and a blood pressure will be recorded. Angina pectoris at any point during these tests will be an indication that the test needs to be stopped and the heart rate will be allowed to return to normal.

This assessment will be undertaken twice during this first visit, once with MPP on and once with MPP off in random order.

Following these echocardiographic assessments (which will occur at rest on the echo couch), patients will undergo a peak walk test on the treadmill during which peak oxygen consumption (a cardiopulmonary exercise test) will be assessed. Prior to this test, the pacemaker heart rate programming will be optimised in line with previous data, and MPP will be either activated or left off in random order with allocation carried out in a double-blind fashion. Participants will be invited back at one week (7 weeks after the implant procedure) for a second exercise test for the second arm (MPP off or on).

Images will be stored for offline analysis and governance purposes. Pacemaker devices will be set to usual programming modes at the end of each visit.

Six months after the device implant:

At around 6 months after the initial implant, the above protocol will be repeated with two echocardiograms and one exercise test at the first visit and one exercise test one week later. At one of these 6-month visits, patients will be asked to complete two quality of questionnaires (Minnestoa Living with Heart Failure and the EQ5D-5L).

Long term assessment (phase 2):

At six months, patients will be invited to continue into a second stage during which MPP will be randomly programmed on or left off. This will be a double-blind, randomised, parallel cohort study. Participants will come back at a further 6 months (12 months after implant) for a final visit which will include echocardiography and a treadmill test and also complete the two quality of life questionnaires. At this point, unless there is clear evidence of benefit of MPP, we will decide to turn off this programming mode in those that were randomised to 'MPP-on', or on in those randomised to 'MPP-off'. This will be based upon individual assessment until the results of the entire study are known.

Data analysis plan A measure of contractility will be collected at each heart rate interval. These can be plotted against heart rate for each patient to achieve three novel variables per patient (peak contractility, heart rate for peak contractility and the slope of the FFR). The study aims to determine whether these three variables change over time following CRT implantation, and whether they are influenced by MPP.

These comparison projects and the randomised placebo-controlled trial are exploratory and feasibility studies respectively. The sample size for the former will be reviewed after the first 10 patients are enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic heart failure due to left ventricular systolic dysfunction (LVEF<35%)
2. Due to (or just undergone) undergo CRT implantation
3. Able to perform a peak exercise test
4. Willing and able to give informed consent

Exclusion Criteria:

1. Atrial fibrillation
2. Angina pectoris symptoms limiting exercise tolerance
3. Unstable heart failure symptoms (medical therapy changes in last three months
4. Poor imaging quality such that analysis is unreliable
5. Calcium channel blockers (CCBs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Force frequency curve (phase 1) | Acute - cross-over phase at 6 weeks
  Contractility curve over heart rate range

SECONDARY OUTCOMES:
Quality of life (MLWHF) | From 6 months to 12 months following implant
  Minnesota Living with Heart Failure
Quality of life (EQ5D-5L) | From 6 months to 12 months following implant
  EQ5D-5L
Treadmill walk time (phase 2) | From 6 months to 12 months following implant - chronic parallel group phase
  Time to exhaustion on a treadmill
Force frequency curve (phase 1) | Acute - cross-over phase at 6 months
  Contractility curve over heart rate range

OTHER OUTCOMES:
Battery longevity after 6 months of MPP versus usual pacing | From 6 months to 12 months following implant
  As predicted by device

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Witte, MD, Principal Investigator — University of Leeds
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Not yet planned